CLINICAL TRIAL: NCT01418729
Title: Phase-II, Multicenter, Randomized, Double-Blind, Parallel-Group Trial to Compare the Efficacy and Safety of Sorafenib Plus Pravastatin Against Sorafenib Plus Placebo in Patients With Advanced Hepatocarcinoma
Brief Title: Efficacy and Safety Study of Sorafenib Plus Pravastatin to Treat Advanced Hepatocarcinoma
Acronym: ESTAHEP-2010
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Donostia (Other)
Collaborators: INSTITUTO BIODONOSTIA (Unknown)
Responsible Party: Principal Investigator, Juan I. Arenas Ruiz-Tapiador, MD. PHD, Hospital Donostia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESTAHEP-2010; 2010-024421-21 (EudraCT Number)
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Advanced Hepatocarcinoma
MeSH Terms: interventions — Pravastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib plus Pravastatin (Active Comparator): The treatment received will be sorafenib 400 mg/12 h + pravastatin 40 mg/24 h.
  Interventions: Drug: Pravastatin
- Sorafenib plus Placebo (Placebo Comparator): The treatment received will be sorafenib 400 mg/12 h + placebo/24 h.
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — Treatment:
  Patients will be randomized in two groups, A and B:
  * Control Group (A ≡ 1): Patients will receive treatment with sorafenib 400 mg/12 h + placebo/24 h.
  * Experimental Group (B ≡ 2): The treatment received will be sorafenib 400 mg/12 h + pravastatin 40 mg/24 h.

SUMMARY:
The purpose of this study is to evaluate the overall survival (OS) in order to assess the efficacy and safety of pravastatin as adjuvant treatment to sorafenib.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been diagnosed with advanced hepatocarcinoma (HCC), confirmed histologically or with non-invasive criteria, according to the clinical practice guidelines by the American Association for the Study of Liver Diseases (AASLD) during a maximum period of 15 days prior to the baseline visit.
* Males and females, over 18 years of age.
* Patients who have not previously received treatment with sorafenib.
* Have an ECOG ≤ 2.
* Liver function: Child A and B7.
* Life expectancy greater than 12 weeks.
* Adequate kidney function: serum creatinine concentration less than or equal to 1.5 times the upper limit of normal (ULN).
* Sign the written informed consent before starting any procedure, including randomization.

Exclusion Criteria:

* Patients who routinely (more than 3 times a week) take some sort of statin.
* Patients with hypersensitivity to statins.
* Pregnant or breastfeeding women.
* Peripheral neuropathy: grade 2 or higher
* Patients who have been diagnosed, within the previous 5 years, with another type of tumor, except for non-melanoma skin cancer, or in situ carcinoma of the cervix or the urinary bladder.
* Patients receiving chemotherapy or radiotherapy for another type of tumor.
* Patients with heart failure greater than NYHA grade II, hypertension that is uncontrolled with medication, uncontrolled arrhythmias or AMI within the previous six months.
* A history of perforation or hemorrhage due to a gastroduodenal ulcus within the last month.
* Greater hemorrhagic diseases.
* Asthmatic patients uncontrolled with medication.
* Any other contraindication associated to the use of statins.
* Physical or psychological inability to participate in the trial.
* Treatment with another investigational drug or participation in another clinical trial within 6 months prior to inclusion in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Overall survival | 18 months
  To evaluate the overall survival (OS) in order to assess the efficacy and safety of pravastatin as adjuvant treatment to sorafenib.

SECONDARY OUTCOMES:
Time to progression | 18 months
  To evaluate the time to progression (TTP).
time to symptomatic progression (TTSP). | 18 months
  To evaluate the time to symptomatic progression (TTSP).

CONTACTS AND LOCATIONS:
Overall Officials: Juan I Arenas, MD,PHD, Study Chair — Hospital Donostia; Javier Bustamante Scheneider, MD, Principal Investigator — Hospital de Cruces; Trinidad Serrano Aullo, MD, PHD, Principal Investigator — Hospital Clínico Universitario Lozano Blesa; Mercedes Iñarrairaegui Bastarrica, MD, Principal Investigator — Clínica Universitaria de Navarra; Sonia Blanco Sampascual, MD, Principal Investigator — Hospital de Basurto; Maria Varela, MD, PHD, Principal Investigator — Hospital Central de Asturias; Oscar Nuñez, MD, Principal Investigator — Hospital Infanta Sofia
Locations (1):
- Hospital Donostia, Instituto Biodonostia, Donostia / San Sebastian, Gipuzkoa, Spain

REFERENCES:
- See also: Related Info — http://www.biodonostia.org